CLINICAL TRIAL: NCT04445948
Title: Study the Efficacy of Lactoferrin in Helicobacter Pylori Eradication Either With Standard Triple Therapy or Sequential Therapy in Egyptian Patients
Brief Title: Lactoferrin in Helicobacter Pylori Eradication Either With Standard Triple Therapy or Sequential Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Collaborators: University of Alexandria (Other)
Responsible Party: Principal Investigator, Sameh A. Lashen, Associate Professor of Internal Medicine., Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0304432
Record Dates: First submitted 2020-06-21; First posted 2020-06-24 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Helicobacter Pylori Infection
Keywords: H.pylori; Lactoferrin; triple therapy
MeSH Terms: interventions — Esomeprazole; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Triple Therapy (Active Comparator): Received triple therapy in the form of esomeprazole 40 milligrams tablets once daily 30 minutes before breakfast plus amoxicillin 1 gram tablets twice daily and clarithromycin 500 milligrams tablets twice daily after meal for 14 days.
  Interventions: Drug: Esomeprazole 40 milligrams Oral Tablet; Drug: Amoxicillin 1000 milligrams tablets; Drug: Clarithromycin 500 milligrams Tablets
- Sequential Therapy (Active Comparator): Received the sequential therapy in the form of esomeprazole 40 milligrams tablets once daily 30 minutes before breakfast plus amoxicillin 1 g tablets twice daily for 5 days, then esomeprazole 40 milligrams tablets once daily 30 minutes before breakfast plus metronidazole 500 milligrams tablets twice daily plus clarithromycin 500 milligrams tablets twice daily after meal for another 10 days.
  Interventions: Drug: Esomeprazole 40 milligrams Oral Tablet; Drug: Amoxicillin 1000 milligrams tablets; Drug: Clarithromycin 500 milligrams Tablets; Drug: MetroNIDAZOLE 500 milligrams Oral Tablet
- Triple Therapy plus Lactoferrin (Active Comparator): Received triple therapy in the form of esomeprazole 40 milligrams tablets once daily 30 minutes before breakfast plus amoxicillin 1 gram tablets twice daily and clarithromycin 500 milligrams tablets twice daily after meal for 14 days. in addition to 200 milligrams of bovine lactoferrin sachets twice daily 30 minutes after breakfast and dinner for 14 days.
  Interventions: Drug: Esomeprazole 40 milligrams Oral Tablet; Drug: Amoxicillin 1000 milligrams tablets; Drug: Clarithromycin 500 milligrams Tablets; Drug: Lactoferrin Bovine sachets 200 milligrams
- Sequential Therapy plus Lactoferrin (Active Comparator): Received the sequential therapy in the form of esomeprazole 40 milligrams once daily 30 minutes before breakfast plus amoxicillin 1 gram twice daily for 5 days, then esomeprazole 40 mg once daily 30 minutes before breakfast plus metronidazole 500 milligrams twice daily plus clarithromycin 500 milligrams twice daily after meal for another 10 days in addition to 200 milligrams of bovine lactoferrin sachets twice daily 30 minutes after breakfast and dinner throughout the 15 days.
  Interventions: Drug: Esomeprazole 40 milligrams Oral Tablet; Drug: Amoxicillin 1000 milligrams tablets; Drug: Clarithromycin 500 milligrams Tablets; Drug: MetroNIDAZOLE 500 milligrams Oral Tablet; Drug: Lactoferrin Bovine sachets 200 milligrams

INTERVENTIONS:
Drug: Esomeprazole 40 milligrams Oral Tablet — Proton Pump inhibitor
  Other Names: Nexium; Esompex
Drug: Amoxicillin 1000 milligrams tablets — Penicillin derivative antibiotic
  Other Names: Amoxil; Amoxicillin
Drug: Clarithromycin 500 milligrams Tablets — Macrolide antibiotic
  Other Names: Klacid; Klarithro
Drug: MetroNIDAZOLE 500 milligrams Oral Tablet — Antiprotozoal
  Other Names: Amrizole; Flagyle
  Arms: Sequential Therapy; Sequential Therapy plus Lactoferrin
Drug: Lactoferrin Bovine sachets 200 milligrams — a protein found naturally in milk from humans and cows
  Other Names: Pravotin
  Arms: Sequential Therapy plus Lactoferrin; Triple Therapy plus Lactoferrin

SUMMARY:
The investigators aim at evaluating the efficacy of bovine lactoferrin addition to H. Pylori eradication regimens. 400 randomly distributed participants will be assigned to one of four treatment regimens of H. Pylori (standard triple therapy, standard triple therapy plus bovine lactoferrin, sequential therapy, or sequential therapy plus bovine lactoferrin), and eradication rates will be evaluated among the four groups.

DETAILED DESCRIPTION:
the study included 400 patients recruited from Gastroenterology as well as general internal medicine clinic at Internal Medicine department, Faculty of Medicine, University of Alexandria, Egypt. After initial evaluation, every participant was randomly assigned to one of four equal treatment regimens (using simple randomization, 100 patients for each regimen) All included participant subjected to evaluation as regards demographic parameters, current status of smoking, history of dyspepsia, epigastric pain, heartburn, melena, hematemesis, nauseas / vomiting, weight loss, and dysphagia.

The diagnosis of H. Pylori infection was based on positivity of H. Pylori stool antigen (HpSAg) in patients who were not indicated for upper endoscopic study / or rapid urease test during esophagogastroduodenoscopy (EGD).

The HpSAg enzyme-linked immunoassay was read spectrophotometrically at 450 nm and the results are recorded as negative if the optical density (O.D.) is <0.14, positive if O.D. ≥0.16, and equivocal for any values ≥0.14 and <0.16.

Upper endoscopy was done to all patients above 45 years of age or patients with alarming symptoms (melena, hematemesis, weight loss, and dysphagia) or family history of gastric cancer.

Rapid urease test was done during EGD as an invasive tool for diagnosis of H.Pylori infection.

After diagnosis, patients were randomly assigned as following:

group (A) received the triple therapy for 2 weeks in the form of esomeprazole 40 milligrams once daily 30 minutes before breakfast plus amoxicillin 1 gram twice daily and clarithromycin 500 milligrams twice daily after meal; group (B) received the sequential therapy in the form of esomeprazole 40 milligrams once daily 30 minutes before breakfast plus amoxicillin 1 gram twice daily for 5 days and then esomeprazole 40 milligrams once daily 30 minutes before breakfast plus metronidazole 500 milligrams twice daily and clarithromycin 500 milligrams twice daily after meal for 10 days; group (C) received the triple therapy for 2 weeks in addition to 200 milligrams of commercially available bovine lactoferrin twice daily 30 minutes after breakfast and dinner for 14 days; group (D) received the sequential therapy in addition to 200 milligrams of commercially available bovine lactoferrin twice daily 30 minutes after breakfast and dinner for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Age group 18-60 years,
* Positive H. Pylori test (Stool antigen / or rapid urease test)

Exclusion Criteria:

* The use of proton pump inhibitor , H2-receptor antagonist, bismuth preparation and antibiotics at least 2 weeks before enrollment,
* prior eradication treatment,
* History of gastrectomy,
* Equivocal H. pylori stool antigen (HpSAg) results,
* Severe hepatic (Child Pugh class B or C) or renal diseases (eGFR < 60 ml/min/1.73 m^2),
* Any form of malignancy,
* Proven allergy to clarithromycin, or Penicillin,
* Pregnant or lactating females.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2019-11-30 (Actual); Primary Completion 2020-06-21 (Actual); Study Completion 2020-06-21 (Actual)

PRIMARY OUTCOMES:
H. Pylori eradication rate | evaluated 28 days after last dose of treatment
  H. Pylori eradication rate among the four groups as evaluated by negativity of H. Pylori stool antigen

CONTACTS AND LOCATIONS:
Overall Officials: Sameh A Lashen, MD(PhD), Principal Investigator — University of Alexandria
Locations (1):
- Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No
data confidentiality will be preserved